CLINICAL TRIAL: NCT06719167
Title: Residential Group and Individual Trauma Informed Stabilization Therapy for Adult Survivors of Childhood Trauma
Brief Title: A Pilot Research Project on Outcome of Trauma Informed Stabilization Treatment (TIST) for Adults with Complex Trauma Symptoms After Childhood Trauma, At the Department of Trauma Treatment, Modum Bad, Norway
Status: Enrolling by invitation | Type: Observational
Sponsor: Modum Bad (Other)
Responsible Party: Sponsor
Other Study IDs: TIST pilot project
Record Dates: First submitted 2024-11-20; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: PTSD and Trauma-related Symptoms; PTSD
Keywords: complex PTSD; childhood trauma; TIST; group treatment; affect regulation; mindfulness; self compassion
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment: All group and individual therapy will be in line with the Trauma Informed Stabilization Treatment (TIST) model, developed by dr Janina Fisher. Patients will be admitted for in-patient pre-planned treatment over 11 weeks in an open door psychiatric hospital. Patients will be summoned for 6 day follow-up 8 months after discharge.
  Interventions: Behavioral: Psychoterapy

INTERVENTIONS:
Behavioral: Psychoterapy — During 11 weeks admission the programme will include group sessions using different modalities (psychoeducation videos, live psychoeducation groups, expressive arts therapy, equine facilitated therapy, mindfulness and discussion groups) all using TIST methodology. Parallell individual therapy with therapist (psychologist or psychiatrist) and milieu therapist. All therapists will be trained minimum in TIST level 1 and recieve supervision from an expert TIST therapist.
  Other Names: TIST; Trauma Informed Stabilization Treatment

SUMMARY:
The purpose of the study is to examine the effects of residential group and individual Trauma Informed Stabilization Treatment (TIST) for complex symptoms in adult survivors of childhood trauma in a naturalistic observational study.

DETAILED DESCRIPTION:
Adult survivors of childhood trauma have complex and diverse symptom profiles. The aim of the study is to examine the effects of theTrauma Informed Stabilization Treatment (TIST) model, developed by dr Janina Fisher, in adult survivors of childhood trauma.

32 patients will be recruited from referrals to an residential open door trauma clinic in Norway, Modum Bad. Patients will be admitted for in-patient pre-planned treatment over 11 weeks - consisting of individual therapy and group therapy using different modalities, all within the TIST approach and framework. Patients will be summoned for 6 day follow-up 8 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years
* Complex symptom presentations connected to childhood trauma
* All patients will have undergone outpatient therapy with insufficient effect
* Most included patients will have a diagnosis of complex PTSD (diagnosed by M.I.N.I. and clinical evaluation)
* Patients may have diagnosis of unspecified dissociative disorder, personality disorders, depression and other comorbidity.

Exclusion criteria:

* Dissociative identitiy disorder
* Ongoing psychosis
* Ongoing drug addiction
* Very disturbed group function
* Ongoing life crisis
* Mental disability
* Acute suicidality
* Ongoing severe self harm
* Patients with complex dissociative disorders and patients eligible for exposure therapy will be referred to/prioritized for other treatment programmes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from referrals to the clinic after assessment of eligibilty criteria.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Difficulties in emotion regulation scale (DERS) | Week 0 (Admission), week 11-12 (discharge) and 8 months follow up
  Difficulties in emotion regulation scale, scale and subscales
Five facet mindfulness questionnaire (FFMQ) | Week 0 (Admission), week 11-12 (discharge) and 8 months follow up
  Five facet mindfulness questionnaire, all subscales
Self-compassion scale long form (SCS-LF) | Week 0 (Admission), week 11-12 (discharge) and 8 months follow up
  Self-compassion scale long form, scale and subscales
PTSD checklist for DSM-5 (PCL-5) | Week 0 (Admission), week 11-12 (discharge) and 8 months follow up
  PTSD checklist for DSM-5, scale and subscales
International trauma questionnaire (ITQ) | Week 0 (Admission), week 11-12 (discharge) and 8 months follow up
  International trauma questionnaire, scale and subscales

SECONDARY OUTCOMES:
Patient health questionnaire 9 (PHQ-9) | Week 0 (Admission), week 11-12 (discharge) and 8 months follow up
  Patient health questionnaire 9
Quality of life | Week 0 (Admission), week 11-12 (discharge) and 8 months follow up
  Self report on scale of 0-10

CONTACTS AND LOCATIONS:
Locations (1):
- Modum Bad, Vikersund, Buskerud, Norway

IPD SHARING:
Plan to Share IPD: Undecided